CLINICAL TRIAL: NCT06119568
Title: HYbrid RObotic Surgery in Partial, Radical Nephrectomy and Prostatectomy (HYROS-PRnP)
Brief Title: Safety and Performance Assessment of a First Four Arms on Demand Open Robotic Solution for Assisted PN, RN and RP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rob Surgical Systems S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PL-PR01-076
Record Dates: First submitted 2023-10-27; First posted 2023-11-07 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-01

CONDITIONS: Nephrectomy; Prostatectomy
Keywords: Radical nephrectomy; Partial nephrectomy; Radical prostatectomy; Lymphadenectomy; Lysis of adhesion; Robotic surgery; Minimal invasive surgery; Robotic minimal invasive surgery; Urology
MeSH Terms: interventions — Nephrectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients surgically treated with Bitrack System and ESE/ NESE instruments and accessories (Experimental)
  Interventions: Device: Robot assisted laparoscopic Radical/simple nephrectomy (RN), Partial nephrectomy (PN) or Radical Prostatectomy (RP).

INTERVENTIONS:
Device: Robot assisted laparoscopic Radical/simple nephrectomy (RN), Partial nephrectomy (PN) or Radical Prostatectomy (RP). — Three different surgery interventions: 1. Radical Nephrectomy: Complete remove of the kidney; 2. Partial Nephrectomy: Partial remove of a section in the kidney. 3. Radical Prostatectomy: Complete remote of the prostate gland. During each of these procedures removal of regional lymph nodes (lymphadenectomy) and lysis of abdominal lesions may be performed according to patient medical condition and/or surgeon criteria.

SUMMARY:
The purpose of this clinical investigation is to evaluate the safety and performance of the Bitrack System and its corresponding ElectroSurgical Endoscopic (ESE) instruments and Non-ElectroSurgical Endoscopic (NESE) instruments and accessories in patients with the indication of a robot assisted laparoscopic Radical Nephrectomy (RN), Partial Nephrectomy (PN) or Radical Prostatectomy (RP), as applicable. HYROS-PRnP is a confirmatory study in which the hypothesis of the primary endpoint is that the ESE/NESE instruments perform as intended when controlled by Bitrack System which operates exclusively under surgeon's orders. The study shall refer to safety and performance of Bitrack System together with its accessories and corresponding ESE/NESE instruments. This study includes the data collected up to 30 days post-surgery and provides the evidence that the tested medical devices fulfill the GSPR.

DETAILED DESCRIPTION:
The Bitrack System is first 4-arms on demand open robotic platform indicated to be used during general abdominal laparoscopic urologic surgical procedures. This robot is intended to assist in the accurate control of endoscopic instruments and accessories for visualization and endoscopic manipulation.

The HYROS-PRnP clinical investigation will be conducted as a single-center, with a single arm, open-label, and non-randomized design, that will include 15 patients. This clinical investigation aims to evaluate the safety and performance of the Bitrack System in patients indicated with robotic-assisted laparoscopic Radical nephrectomy, Partial nephrectomy or Radical Prostatectomy surgeries.

The planned visits for this clinical investigation are baseline (includes Screening, baseline visit, and Informed consent), procedure, discharge, 14-Days Follow-up visit, and 30-Days Follow-up visit (remote). The clinical investigation will include adult subjects (between 18 and 90 years old) who have been scheduled for laparoscopic Radical Nephrectomy. Partial Nephrectomy or Radical Prostatectomy. The total duration of the clinical investigation is expected to be 4 months, consisting of approximately 3 months of enrollment plus 1 month of follow-up. The end of the clinical investigation will occur when the last visit of the last enrolled subject is completed.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects between 18 and 90 years old who have provided written informed consent prior to any clinical investigation related procedures.
2. Subjects who have been scheduled for a laparoscopic Radical/simple Nephrectomy surgery, laparoscopic Partial Nephrectomy or laparoscopic Radical Prostatectomy following the surgeon criteria.
3. Ability and willingness to comply with all study requirements to be evaluated for each study visit.

Exclusion Criteria:

1. Pregnant or breastfeeding women at the time of the surgery.
2. Subjects with severe concomitant illness that, at PI´s discretion, increases risk of therapeutic interventions or that have been submitted to multiple prior surgeries.
3. Subjects admitted to the hospital due to an emergency situation.
4. Subjects with untreated active infection.
5. Subject with known allergy to some of the device components (i.e., stainless steel, etc.)
6. Subjects not suitable to undergo MIS/MIRS, according to medical criteria.
7. Subjects with life expectancy inferior to 3 months.
8. Subjects with a BMI ≥ 40.
9. Subjects with any contraindication for the use of the Bitrack System and the ESE/NESE instruments, as specified in the Instructions For Use.
10. Subjects with abuses of active substances or with uncontrolled psychiatric disorders.
11. Subjects with severe cardiopulmonary or coronary artery disease, bleeding disorders or that have been submitted to multiple prior operations.
12. Subjects scheduled for surgeries intended to be in direct contact with the heart, the central circulatory system or the central nervous system.
13. Inability to adhere to study-related procedures.
14. Subjects who participate in another trial which may affect the outcome data on this study or the ability to complete the follow up requirements.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
Lack of occurrence of a SAE related to the use of the medical devices under investigation during the intervention | During the procedure
  Evaluation of Bitrack System to assist in the accurate control of its compatible ESE/NESE instruments, during the intervention without causing any particular SAE related to the use of the medical devices under investigation.
Performance | During the procedure
  Assessment with a "Surgeon performance scale" to confirm that the Bitrack system and ESE/NESE instruments perform as intended during the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Lluís Peri Cusí, MD, Principal Investigator — Urology Department, Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain